CLINICAL TRIAL: NCT02220634
Title: Regadenoson for Acute Vasoreactivity Testing in Pulmonary Hypertension
Acronym: RHINO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left National Jewish Health
Sponsor: National Jewish Health (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-2820
Record Dates: First submitted 2014-05-06; First posted 2014-08-20 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary | interventions — regadenoson

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Regadenoson (Experimental): Intravenous infusion of the A2A agonist regadenoson has a preferential vasodilator effect on pulmonary vasculature that is comparable to iNO, the current gold standard for pulmonary vasoreactivity studies.
  Interventions: Drug: Regadenoson

INTERVENTIONS:
Drug: Regadenoson — Injection for intravenous administration
  Other Names: Lexiscan

SUMMARY:
The purpose of this study is to see if Regadenoson may offer improved ease of use, single dose administration, and better tolerance for testing for pulmonary hypertension than iNO. You will be screened to make sure Regadenoson is safe for you with a clinical evaluation, blood tests, and an ECG.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) is an increase of blood pressure in the pulmonary vascular system that could cause shortness of breath, dizziness, leg swelling and heart failure. .

The diagnosis of PH requires confirmation of elevated pulmonary pressures.. Right heart catheterization (RHC) is a procedure to determine the diagnosis of PH. .

This research study is looking at the effect of intravenous infusion of the medication Regadenoson on pulmonary vasodilator response compared to the inhaled nitric oxide (iNO) response. iNO is the current standard of care practice.

The purpose of this study is to see if Regadenoson may offer improved ease of use, single dose administration, and better tolerance for testing for pulmonary hypertension than iNO. You will be screened to make sure Regadenoson is safe for you with a clinical evaluation, blood tests, and an ECG.

You will be asked to sign this informed consent form. Then, you will undergo right heart catheterization as part of your clinical care. Those who are positive for pulmonary hypertension will then undergo Regadenoson infusion and a inhaled iNO. Prior to the infusion, subjects will be asked if they have had in the last 12 hours any caffeine-containing foods or beverages, caffeine-containing medications such as theophylline 12 hours prior. Vital sign measurements will be taken to measure your heart. For those subjects that have low heart volume they will be given 500 cc of normal saline in their IV. Vital sign measurements will be taken again to make sure your heart volume is in the normal range. The doctor will administer Regadenoson 0.4 mg intravenously and this will cause your heart rate to increase. The doctor will be taking heart measurements 90 seconds, 5 minutes, 10 minutes, and 20 minutes after administration. Approximately 30 minutes after the Regadenoson has been administered you will be given iNO by facemask for 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old
2. Diagnosis of RHC-proven PH

   * Mean pulmonary artery pressure (mPAP) > 25 mmHg
   * Pulmonary vascular resistance (PVR) > 3 woods units
   * Pulmonary capillary wedge pressure (PCWP) < 15 mmHg).

Exclusion Criteria:

1. Second- or third-degree AV block or sinus node dysfunction
2. Known hypersensitivity to adenosine or regadenoson
3. Systolic blood pressure < 90mm Hg
4. Active bronchospasm
5. Autonomic dysfunction as defined by prior diagnosis of:

   * Postural Orthostatic Tachycardia Syndrome (POTS)
   * Neurocardiogenic Syncope (NCS)
   * Neurally Mediated Hypotension (NMH)
   * Vasovagal Syncope
6. Hypovolemia
7. > 40% Left main coronary stenosis
8. Moderate or > valvular stenosis
9. Pericarditis/pericardial effusions
10. > 70% carotid artery stenosis
11. Positive urine pregnancy test

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-08; Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Number of people | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Brett E Fenster, MD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Health, Denver, Colorado, United States